CLINICAL TRIAL: NCT02865837
Title: Effect of Bladder Distension on Organs at Risk Doses in PDR 3D Image-guided Brachytherapy of Cervical Cancer
Brief Title: Effect of Bladder Distension on Dosimetry in Brachytherapy of Cervical Cancer
Acronym: VESICOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Cancérologie de Lorraine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2015-A00923-46
Record Dates: First submitted 2016-07-04; First posted 2016-08-15 (Estimated); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Cervical Cancer
Keywords: Brachytherapy; Organs at Risk; Bladder volume; Cervical cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Brachytherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ARM 1 (Experimental)
  Interventions: Other: brachytherapy

INTERVENTIONS:
Other: brachytherapy — The brachytherapy applicator and a urinary catheter are set up in the operating room under general anesthesia.
  Then, an MRI (or a scanner if contra-indication) is performed after a bladder filling with 120cc of normal saline solution and urinary catheter clamping.
  Right after, a scanner is performed with urinary catheter declamping and emptied bladder.
  Delineation of CTVs and organs at risk (bladder, rectum, sigmoid, small bowel), and dosimetric optimisation are made on study with filled bladder.
  Then, organs at risk are delineated on the study with emptied bladder. The prior dosimetry is reset on this study and organs at risk doses are compared.

SUMMARY:
The purpose of this study is to compare, for each patient, dosimetry of organs at risk (bladder, rectum, sigmoid, small bowel) in two bladder distension procedures (emptied by a urinary catheter or filled with 120cc) during PDR 3D image-guided brachytherapy of cervical cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age > or = 18 years old
* with a cervical cancer histologically proven (squamous cell carcinoma, adenocarcinoma and neuroendocrine cell carcinoma)
* Utero-vaginal brachytherapy indications::

  * Stage 1B1: brachytherapy before surgery
  * Stages IB2 to IIIB: after pelvic radiotherapy (45Gy/25 fractions/5 weeks) with or without concomitant chemotherapy
* Ability to provide an informed written consent form
* Patient must be affiliated to a social security system

Exclusion Criteria:

* Age < 18 years old
* History of pelvic radiotherapy
* History of pelvic surgery
* Recent joint prothesis (<3 months)
* Pregnant woman or being breastfeeding
* Patients deprived of liberty or under supervision

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Demonstrate the non inferiority of 3D image-guided brachytherapy with emptied bladder compared to filled bladder for the dose received by the bladder | 1 day
  Difference of the maximum dose received by 2 cm3 bladder (D2cc) between the two conditions: full and empty.

SECONDARY OUTCOMES:
Non-inferiority based on the dose received by the rectum | 1 day
Non-inferiority based on the dose received by the sigmoid | 1 day
Non-inferiority based on the dose received by the small bowel | 1 day
FIGO staging system | 1 day
Body Mass Index | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: RENARD OLDRINI SOPHIE, MD, Principal Investigator — Institut de Cancérologie de Lorraine
Locations (1):
- Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No